CLINICAL TRIAL: NCT00468676
Title: Randomized Trial of Liaison Psychiatry in Primary Care
Brief Title: Nurse-led Case Management for Diabetes and Cardiovascular Disease Patients With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Wayne Katon, Professor, Vice Chair University of Washington, National Institute of Mental Health (NIMH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH041739 (NIH); R01MH041739 (NIH); DSIR 82-SEPC
Record Dates: First submitted 2007-05-01; First posted 2007-05-03 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Depression
Keywords: major Depressive Disorder; Diabetes; Heart Disease
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Diabetes Mellitus; Heart Diseases | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Active Comparator): Treatment as usual
  Interventions: Behavioral: Treatment as usual
- A (Experimental): Case management intervention
  Interventions: Behavioral: Nurse-led case management

INTERVENTIONS:
Behavioral: Nurse-led case management — The case management intervention will entail approximately 10 visits with a trained nurse at the clinic or by telephone. Participants in this group will receive educational materials about how to manage diabetes and/or heart disease and stress or depression. Nurses will also provide guidance and support in managing medications, phone calls to check participants' progress, and assistance in setting personal goals and in managing physical health problems and symptoms of depression or stress.
  Arms: A
Behavioral: Treatment as usual — Participants will attend 10 study visits and receive 4 follow-up phone calls over 24 months. During this time, participants will receive usual care.
  Arms: B

SUMMARY:
This study will evaluate the effectiveness of a nurse-led case management intervention in improving disease control and depression symptoms in adults with diabetes and/or heart disease who are also depressed.

DETAILED DESCRIPTION:
Depression is a serious medical illness that has been associated with increased risk for heart disease and diabetes. Depression may negatively impact aspects of self-care that are required to effectively manage such long-term diseases. In depressed people who have heart disease and/or diabetes, treatment for depression appears to result in only limited improvements in depression symptoms and no improvements in heart disease and diabetes symptoms. An integrated treatment approach may be more effective in improving all three conditions. This study will evaluate the effectiveness of a nurse-led case management intervention in improving disease control and depression symptoms in adults with diabetes and/or heart disease who are also depressed.

Participants in this single-blind study will be randomly assigned to take part in the case management intervention or receive usual care. All participants will attend 5 in-person study evaluation visits and receive 4 follow-up phone calls over 24 months. At each of the study visits, measurements of height, weight, waist size, and blood pressure will be taken. At study evaluations, blood and urine samples will also be taken. Participants will be asked not to eat for 8 hours before providing blood samples at 3 of the visits. During follow-up phone calls participants will answer various questions.

The case management intervention will entail approximately 10 visits with a trained nurse at the clinic or by telephone. Participants in this group will receive educational materials about how to manage diabetes and/or heart disease and stress or depression. Nurses will also provide guidance and support in managing medications, phone calls to check participants' progress, and assistance in setting personal goals and in managing physical health problems and symptoms of depression or stress. Outcomes will be measured at Months 6, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes and/or heart disease
* Poor disease control (defined as an HbA1c level of at least 8.5%, blood pressure greater than 140/90 mm Hg, LDL cholesterol greater than 130 mg/dL)
* Diagnosis of major depressive disorder

Exclusion Criteria:

* History of psychosis
* At high risk for suicide
* Cognitive impairment
* Current alcohol or substance abuse disorder
* Does not own a telephone
* Currently seeking psychiatric care
* Pregnant or breastfeeding
* Currently enrolled in a Group Health Cooperative disease management program
* Terminal illness
* Plans to leave Group Health Cooperative in less than a year
* Does not speak English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2007-05; Primary Completion 2010-10 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne J. Katon, MD, Principal Investigator — University of Washington
Locations (1):
- Group Health Cooperative, Seattle, Washington, United States

REFERENCES:
- [Result] Katon WJ, Lin EH, Von Korff M, Ciechanowski P, Ludman EJ, Young B, Peterson D, Rutter CM, McGregor M, McCulloch D. Collaborative care for patients with depression and chronic illnesses. N Engl J Med. 2010 Dec 30;363(27):2611-20. doi: 10.1056/NEJMoa1003955. PMID 21190455
- [Result] Lin EH, Von Korff M, Ciechanowski P, Peterson D, Ludman EJ, Rutter CM, Oliver M, Young BA, Gensichen J, McGregor M, McCulloch DK, Wagner EH, Katon WJ. Treatment adjustment and medication adherence for complex patients with diabetes, heart disease, and depression: a randomized controlled trial. Ann Fam Med. 2012 Jan-Feb;10(1):6-14. doi: 10.1370/afm.1343. PMID 22230825
- [Result] Von Korff M, Katon WJ, Lin EH, Ciechanowski P, Peterson D, Ludman EJ, Young B, Rutter CM. Functional outcomes of multi-condition collaborative care and successful ageing: results of randomised trial. BMJ. 2011 Nov 10;343:d6612. doi: 10.1136/bmj.d6612. PMID 22074851
- [Result] Katon W, Russo J, Lin EH, Schmittdiel J, Ciechanowski P, Ludman E, Peterson D, Young B, Von Korff M. Cost-effectiveness of a multicondition collaborative care intervention: a randomized controlled trial. Arch Gen Psychiatry. 2012 May;69(5):506-14. doi: 10.1001/archgenpsychiatry.2011.1548. PMID 22566583
- [Derived] Ludman EJ, Peterson D, Katon WJ, Lin EH, Von Korff M, Ciechanowski P, Young B, Gensichen J. Improving confidence for self care in patients with depression and chronic illnesses. Behav Med. 2013;39(1):1-6. doi: 10.1080/08964289.2012.708682. PMID 23398269
- See also: Related Info — http://teamcarehealth.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from may 2007 to october 2009 from 14 primary care clinics of Group Health Cooperative in Washington State
Pre-assignment Details: Exclusion criteria: terminal illness, residence in long-term care facility, bipolar/schizophrenia, mental confusion suggesting dementia, pregnancy/breast-feeding, use of antipsychotic/mood stabilizer med, severe hearing loss, planned bariatric surgery within 3 months, ongoing psychiatric care
Groups:
- Usual Care: Patients in usual care arm were advised to consult with their primary care physician to receive care for depression and for diabetes, coronary artery disease or both. With the patient's permission their primary care physician was notified about their PHQ-9 (Patient Health Questionnaire 9) score of 10 or greater and poor medical disease control. In addition primary care doctors received laboratory results at baseline, 6 and 12 months regarding HbA1c and at baseline and 12 months on fasting LDL
- Care Management Intervention: Case management intervention: patients assigned to care management received intervention visits with a medical nurse supervised weekly by both a psychiatrist and primary care doctor. Nurses provided psychoeducation, motivational interviewing, behavioral activation and problem solving and carefully tracked medications, side effects, PHQ-9 (Patient Health Questionnaire 9) scores and blood pressure and lab results. Using a registry the medical supervisors recommended changes in medications that the nurse communicated to the patient's individual primary care doctor (who wrote all prescriptions). Nurses also worked with the patient to set self care goals regarding health behaviors such as increasing exercise or improving diet
Period: Overall Study
Arm/Group | Usual Care | Care Management Intervention
Started | 108 | 106
Completed | 92 | 94
Not Completed | 16 | 12
Not completed — Lost to Follow-up | 14 | 11
Not completed — Death | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: Patients in usual care arm were advised to consult with their primary care physician to receive care for depression and for diabetes, coronary artery disease or both. With the patient's permission their primary care physician was notified about their PHQ-9 score of 10 or greater and poor medical disease control. In addition primary care doctors received laboratory results at baseline, 6 and 12 months regarding HbA1c and at baseline and 12 months on fasting LDL
- Care Management Intervention: Case management intervention: patients assigned to care management received intervention visits with a medical nurse supervised weekly by both a psychiatrist and primary care doctor. Nurses provided psychoeducation, motivational interviewing, behavioral activation and problem solving and carefully tracked medications, side effects, PHQ-9 scores and blood pressure and lab results. Using a registry the medical supervisors recommended changes in medications that the nurse communicated to the patient's individual primary care doctor (who wrote all prescriptions). Nurses also worked with the patient to set self care goals regarding health behaviors such as increasing exercise or improving diet
- Total: Total of all reporting groups
Arm/Group | Usual Care | Care Management Intervention | Total
Number analyzed (Participants) | 108 | 106 | 214
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 82 | 81 | 163
  >=65 years | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (12.1) | 57.4 (10.5) | 56.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 51 | 111
  Male | 48 | 55 | 103
Region of Enrollment [Number; unit: participants]
  United States | 108 | 106 | 214

OUTCOME MEASURES:

1. Primary Outcome: Combined Effect of Intervention on SCL-20, Systolic Blood Pressure, LDL and HbA1c
Description: A scaled marginal model approach was used to jointly describe the four 12 month outcomes (SCL-20, HbA1c, systolic BP, LDL: all data submitted as Outcome Measures #2-5 below) and allowed use to test for a primary effect of the intervention among outcomes, scaling each outcome by its standard error, so the intervention effects could be interpreted as effect sizes.The model was estimated by iterating between estimation of the covariance associated with the outcomes and generalized-estimating equation estimation of scaled outcomes. Effect size is estimated as Cohen d effect size that was use for the depression outcome is the difference in change from baseline to 12 months in the intervention and usual care groups divided by the pooled base line standard deviation. Thus, a d of 0.25 indicates that one-quarter of a standard deviation separates the two means. Cohen has suggested that an effect size of 0.20 would be considered small, 0.50 medium and 0.80 large.
Time Frame: Baseline to 12 months
Population: This was an intent to treat analysis of the 12 month SCL-20, HbA1c, LDL and systolic blood pressure outcomes
Measure: Number (95% Confidence Interval); unit: unitless
Groups:
- Effect Size of Invervention Group to Standard Care: This was an intent to treat analysis calculating the intervention effect size of the 12 month SCL-20, HbA1c, LDL and systolic blood pressure outcomes combined
Arm/Group | Effect Size of Invervention Group to Standard Care
Number analyzed (Participants) | 214
unitless | -1.57 (0.66) [-2.12 to -1.02]
Statistical Analysis 1: Comparison: Effect Size of Invervention Group to Standard Care; Test type: Superiority or Other; p = .001, Scaled Marginal Model — Significance of the four outcome composite; scaled marginal model parameter = -1.57, 95% CI 2-sided [-2.12 to -1.02], Standard Error of Mean .28 — Intervention group had significantly lower scaled marginal mean scores than usual care

2. Secondary Outcome: Functional Impairment
Description: Disability was measured by the Sheehan Disability scale which measures the extent to which health interferes with social, vocational and familial functioning each on a 0 to 10 Likert scale where 0 is "not at all" and 10 is "extremely". This scale consists of 3 items which are averaged together to create the average disability score, which ranges from 0 to 10.
Time Frame: Measured at Months 6, 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Care Management Intervention
Number analyzed (Participants) | 108 | 106
units on a scale
  6-month follow-up | 4.2 (2.6) | 3.7 (3.2)
  12-month follow-up | 4.5 (2.9) | 3.8 (3.0)
Statistical Analysis 1: Comparison: Usual Care vs Care Management Intervention; Disability outcomes were measured at six and 12 months after randomization using linear regression models adjusted for baseline values. The disability models combined information across time points and were estimated using general estimating equations to account for correlation. All analyses were based on intent to treat principles; Test type: Superiority or Other; p < 0.01, general estimating equations; Slope = 0.01

3. Secondary Outcome: Health Care Costs
Description: Mean total outpatient costs for 2 years post baseline adjusted for age, gender and previous 12 months of outpatient costs
Time Frame: Cumulative outpatient costs over 24 months
Measure: Least Squares Mean (Standard Deviation); unit: US dollars
Arm/Group | Usual Care | Care Management Intervention
Number analyzed (Participants) | 108 | 106
US dollars | 21,513 (9201) | 20,918 (10,419)

4. Primary Outcome: Symptom Checklist-20 Score at Baseline, 6 Months and 12 Months
Description: SCL-20 is a 20 question checklist in which items are averaged to yield a potential score of 0 to 4 with higher scores indicating more severe depression symptoms.
  For the Primary Outcome (Outcome Measure #1 above), a scaled marginal model approach was used to jointly describe the four 12 month outcomes (SCL-20, HbA1c, systolic BP, LDL) and allowed use to test for a primary effect of the intervention among outcomes, scaling each outcome by its standard error, so the intervention effects could be interpreted as effect sizes.
Time Frame: Measured at Baseline, 6 Months, 12 months
Population: This was an intent to treat analysis of the 12 month SCL-20, HbA1c, LDL and systolic blood pressure outcomes
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Care Management Intervention: Case management intervention: patients assigned to care management received intervention visits with a medical nurse supervised weekly by both a psychiatrist and primary care doctor. Nurses provided psycho-education, motivational interviewing, behavioral activation and problem solving and carefully tracked medications, side effects, PHQ-9 (Patient Health Questionnaire 9) scores and blood pressure and lab results. Using a registry the medical supervisors recommended changes in medications that the nurse communicated to the patient's individual primary care doctor (who wrote all prescriptions). Nurses also worked with the patient to set self care goals regarding health behaviors such as increasing exercise or improving diet
Arm/Group | Usual Care | Care Management Intervention
Number analyzed (Participants) | 106 | 105
scores on a scale
  SCL-20 at Baseline | 1.65 (0.60) | 1.74 (0.59)
  SCL-20 at 6 mos | 1.26 (0.72) | 0.84 (0.68)
  SCL-20 at 12 mos | 1.14 (0.66) | 0.83 (0.68)
Statistical Analysis 1: Comparison: Usual Care vs Care Management Intervention; Test type: Superiority or Other; p < 0.001, Generalized-Estimating-Equation Model; Estimated Between Group Difference = -0.41, 95% CI 2-sided [-0.56 to -0.26] — Between Group Difference is the difference in the change from Baseline to 12 month data calculated from a generalized-estimating-equation model predicting a 6- and 12-month outcome

5. Primary Outcome: Systolic Blood Pressure at Baseline, 6 Months and 12 Months
Description: Systolic Blood Pressure was measured at Baseline, 6 months and 12 months
  For the Primary Outcome (Outcome Measure #1 above), a scaled marginal model approach was used to jointly describe the four 12 month outcomes (SCL-20, HbA1c, systolic BP, LDL) and allowed use to test for a primary effect of the intervention among outcomes, scaling each outcome by its standard error, so the intervention effects could be interpreted as effect sizes.
Time Frame: Measured at Baseline, 6 Months, 12 months
Population: This was an intent to treat analysis of the 12 month SCL-20, HbA1c, LDL and systolic blood pressure outcomes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Usual Care | Care Management Intervention
Number analyzed (Participants) | 106 | 105
mmHg
  Systolic Blood Pressure at Baseline | 131.9 (17.0) | 135.7 (18.4)
  Systolic Blood Pressure at 6 months | 133.5 (20.4) | 131.9 (15.2)
  Systolic Blood Pressure at 12 months | 132.3 (17.4) | 131.0 (18.2)
Statistical Analysis 1: Comparison: Usual Care vs Care Management Intervention; Test type: Superiority or Other; Generalized-Estimating-Equation Model; Estimated Between Group Difference = -3.4, 95% CI 2-sided [-6.9 to 0.1] — [estimate comment as in outcome 4, analysis 1]

6. Primary Outcome: LDL Cholesterol at Baseline and 12 Months
Description: LDL Cholesterol was measured at Baseline and 12 months
  For the Primary Outcome (Outcome Measure #1 above), a scaled marginal model approach was used to jointly describe the four 12 month outcomes (SCL-20, HbA1c, systolic BP, LDL) and allowed use to test for a primary effect of the intervention among outcomes, scaling each outcome by its standard error, so the intervention effects could be interpreted as effect sizes.
Time Frame: Measured at Baseline and 12 months
Population: This was an intent to treat analysis of the 12 month SCL-20, HbA1c, LDL and systolic blood pressure outcomes
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Usual Care | Care Management Intervention
Number analyzed (Participants) | 106 | 105
mg/dL
  LDL cholesterol at Baseline | 109.4 (36.7) | 106.8 (35.4)
  LDL cholesterol at 12 months | 101.4 (36.6) | 91.9 (36.7)
Statistical Analysis 1: Comparison: Usual Care vs Care Management Intervention; Test type: Superiority or Other; Regression, Linear; Estimated Between Group Difference = -9.1, 95% CI 2-sided [-17.5 to -0.8] — Between Group Difference is the difference in the change from Baseline to 12 month data calculated from a linear-regression model predicting a 12-month outcome

7. Primary Outcome: Glycated Hemoglobin (HbA1c) at Baseline, 6 Months and 12 Months
Description: Glycated hemoglobin (HbA1c) was measured at Baseline, 6 months and 12 months
  For the Primary Outcome (Outcome Measure #1 above), a scaled marginal model approach was used to jointly describe the four 12 month outcomes (SCL-20, HbA1c, systolic BP, LDL) and allowed use to test for a primary effect of the intervention among outcomes, scaling each outcome by its standard error, so the intervention effects could be interpreted as effect sizes.
Time Frame: Measured at Baseline, 6 months and 12 months
Population: This was an intent to treat analysis of the 12 month SCL-20, HbA1c, LDL and systolic blood pressure outcomes
Measure: Mean (Standard Deviation); unit: percent glycated hemoglobin
Arm/Group | Usual Care | Care Management Intervention
Number analyzed (Participants) | 106 | 105
percent glycated hemoglobin
  Glycated Hemoglobin (HbA1c) at Baseline | 8.04 (1.87) | 8.14 (2.03)
  Glycated Hemoglobin (HbA1c) at 6 months | 7.87 (1.93) | 7.42 (1.32)
  Glycated Hemoglobin (HbA1c) at 12 months | 7.81 (1.90) | 7.33 (1.21)
Statistical Analysis 1: Comparison: Usual Care vs Care Management Intervention; Test type: Superiority or Other; Generalized-Estimating-Equation Model; Estimated Between Group Difference = -0.56, 95% CI 2-sided [-0.85 to -0.27] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Groups:
- Usual Care: Treatment as usual
  Treatment as usual: Participants will attend 10 study visits and receive 4 follow-up phone calls over 24 months. During this time, participants will receive usual care.
- Care Management Intervention: Care management intervention
  Nurse-led case management: The case management intervention will entail approximately 10 visits with a trained nurse at the clinic or by telephone. Participants in this group will receive educational materials about how to manage diabetes and/or heart disease and stress or depression. Nurses will also provide guidance and support in managing medications, phone calls to check participants' progress, and assistance in setting personal goals and in managing physical health problems and symptoms of depression or stress.
Arm/Group | Usual Care | Care Management Intervention
Serious Adverse Events (participants affected / at risk) | 2/108 | 1/106
Other Adverse Events (participants affected / at risk) | 23/106 | 27/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=108) | Care Management Intervention (N=106)
Death (General disorders) | 2 | 1 — Deaths that occurred were not due to the study procedures.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=106) | Care Management Intervention (N=105)
Hosptializations (General disorders) | 23 (23) | 27 (27) — Hospitalizations were not the result of the investigation.

LIMITATIONS AND CAVEATS:
Limitations include the study being completed in one health care system in one geographic area, inadequate power to determine cardiovascular events or rates of hospitalization, potential "spill-over of intervention to usual care patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No